CLINICAL TRIAL: NCT00586274
Title: A Phase I Study Evaluating The Use Of Rft5-Dga To Deplete Alloreactive Cells For Patients With Fanconi Anemia After Haploidentical Stem Cell Transplantation
Brief Title: Use of Rft5-Dga to Deplete Alloreactive Cells for Pts With Fanconi Anemia After Haploidentical SCT
Acronym: RAFHAS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Texas, Southwestern Medical Center at Dallas (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-11428
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: FANCONI ANEMIA
Keywords: Stem Cell Transplant; Anemia; Fanconi
MeSH Terms: conditions — Fanconi Anemia; Anemia | interventions — fludarabine; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD34 selected haploidentical PBSCT (Experimental): CD34 selected haploidentical PBSCT
  Interventions: Procedure: CD34 selected haploidentical PBSCT; Drug: Fludarabine; Biological: T cell infusion; Biological: Campath 1h; Biological: anti-CD45

INTERVENTIONS:
Procedure: CD34 selected haploidentical PBSCT — Infusion of CD34 selected haploidentical PBSCT
Drug: Fludarabine — day -8 through day -4 Fludarabine 30 mg/m^2
Biological: T cell infusion — At least 30 days after the stem cell infusion, patients will be dosed with T cells. This study will begin with a dose of T cells known not to cause GvHD even in haploidentical recipients, even when the T cells administered have not first been allodepleted. Dose escalation will follow a traditional up and down method, but as results become available they will be used to determine subsequent dose levels by the continual reassessment method. Initially, 2 patients will be entered beginning at dose level 1. Each and every patient will receive up to three additional injections of T cells at the same dose, at monthly intervals, provided there is no evidence of grade 2 or higher GVHD, until total T cell numbers are > 1000/ul.
  Dose level -1 (1 x 10^3 T cells/Kg); Dose level 1 (1 x 10^4 T cells/Kg); Dose level 2 (1 x 10^5 T cells/Kg); Dose level 3 (1 x 10^6 T cells/Kg); Dose level 4 (5 x 10^6 T cells/Kg)
Biological: Campath 1h — 10 mg iv over 4 hours day-8 through day-6
Biological: anti-CD45 — anti-CD45 400 ug/kg over 6 hours day -5 through day -2

SUMMARY:
While stem cell transplantation has proven an effective means of treating a wide variety of diseases involving hematopoietic stem cells and their progeny, a shortage of donors has proved a major impediment to the widest application of the approach. Until recently, only MHC identical donors could be used with safety. Such donors were originally siblings or other closely related family members. Over the past decade, the growth of allogeneic donor panels has allowed transplantation with stem cells obtained from a volunteer donor panel.

While it is now possible to obtain HLA identical unrelated donor stem cells for approximately 75% of individuals of Northern European backgrounds, the situation for most other ethnic groups is much less satisfactory. Even when a matched donor can be found, the elapsed time between commencing the search and collecting the stem cells usually exceeds three months, a delay that may doom many of the neediest patients. Hence there has been considerable interest in making use of HLA haploidentical family donors. Most individuals have a first-degree relative who would be suitable for such protocols. Fanconi anemia (FA) is an autosomal recessive disorder characterized by the development of progressive aplastic anemia usually evident by about age seven years and often associated with various diverse congenital anomalies such as short stature, microcephaly, radial anomalies, horseshoe kidney, and cafe au lait spots.

This study will determine the number of donor lymphocytes that can be given to recipients of haploidentical stem cell transplants with Fanconi anemia after depletion of recipient-reactive T lymphocytes by ex-vivo treatment with a fixed dose of RFT5-dgA immunotoxin, and will result in a rate of Grade III/IV GVHD of < / = 25%.

DETAILED DESCRIPTION:
Patients will have received a haplo-identical stem cell transplant on our on-going study "CD45 (YTH-24 and YTH-54) and CD52 (Campath 1H) Monoclonal Antibody Conditioning Regimen for Allogeneic Donor Stem Cell Transplantation of Patients with Fanconi Anemia" (H-9938 IND# 7233) and will become eligible to receive allodepleted T Cells following engraftment. What follows is a summary of the treatment plan including initial transplant phase as well as generation and infusion of allodepleted T cells.

Preparative Regimen for Patients with Fanconi Anemia:

The study will be open to patients who received a haploidentical PBSCT on the MAFIA protocol and for patients who failed to engraft and receive a second haploidentical transplants with alternate conditioning consisting of ATG, Fludarabine, TBI (450cGY single dose) and Cytoxan.

In Outline MAFIA conditioning (primary conditioning regimen)

Day 8 Campath 1H 10mg iv over 4hr Fludarabine 30 mg/m2 7 Campath 1H 10mg iv over 4hr Fludarabine 30 mg/m2 6 Campath 1H 10mg iv over 4hr Fludarabine 30 mg/m2 5 YTH 24/54 400ug/kg over 6 hr Fludarabine 30 mg/m2

* 4 YTH 24/54 400ug/kg over 6 hr Fludarabine 30 mg/m2
* 3 YTH 24/54 400ug/kg over 6 hr
* 2 YTH 24/54 400ug/kg over 6 hr
* 1 Rest
* 0 CD34-selected PBSC infusion

Stem Cell Infusion: One day after the completion of pretransplant conditioning therapy (day 0), CD34+ cells will be infused through a central venous catheter as outlined in CAGT SOPs.

This study will begin with a dose of T cells known not to cause GvHD even in haploidentical recipients, even when the T cells administered have not first been allodepleted. Dose escalation will follow a traditional up and down method, but as results become available they will be used to determine subsequent dose levels by the continual reassessment method. Initially, 2 patients will be entered beginning at dose level 1. Each and every patient will receive up to three additional injections of T cells at the same dose, at monthly intervals, provided there is no evidence of grade 2 or higher GVHD, until total T cell numbers are > 1000/ul.

Dose level -1 (1 x 10^3 T cells/Kg); Dose level 1 (1 x 10^4 T cells/Kg); Dose level 2 (1 x 10^5 T cells/Kg); Dose level 3 (1 x 10^6 T cells/Kg); Dose level 4 (5 x 10^6 T cells/Kg)

ELIGIBILITY:
Inclusion Criteria:

* At the time of eligibility for infusion of allodepleted T -cells patients must satisfy the criteria below:
* Patients with Fanconi anemia of all ages with severe aplasia (as evidenced by hypocellular bone marrow) who lack a suitable conventional related (i.e. 5/6 or 6/6 related) or 5/6 or 6/6 unrelated donor with at least 2 out of 3 of the following: a) ANC < 500/mm3, b) reticulocytes < 1% c) platelets < 50,000/mm3
* Diagnosis of Fanconi anemia confirmed by studies of peripheral blood or bone marrow sensitivity to mitomycinC or DEB prior to stem cell transplant. Have received a related haploidentical CD34-selected peripheral blood stem cell transplant with evidence of a full or partial hematopoietic donor chimerism (> 50%) in the peripheral blood.

Exclusion Criteria:

* Patients with a life expectancy (< 6 weeks) limited by diseases other than FA
* Patients with active GVHD > / = Grade II
* Patients with severe renal disease (i.e. creatinine greater than 3 X normal for age)
* Patients with severe hepatic disease (direct bilirubin greater than 3ug/dl or SGPT greater than 500ug/dl)
* Patients with a severe intercurrent infection
* Lansky scale < 60 or Karnofsky < 60

Max Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2002-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Determine # of donor lymphocytes that can be given to recipients of haplo-SCT with FA after depletion of recipient-reactive T lymphocytes by ex-vivo tx with a fixed dose of RFT5-dgA immunotoxin, and will result in Grade III/IV GVHD of < / = 25%. | 1 yr

SECONDARY OUTCOMES:
To analyze immune reconstitution in these patients. | 1 yr
To measure their overall and disease free survival, at 100 days and at 1 year after transplant. | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Brenner, MB, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas